CLINICAL TRIAL: NCT05471713
Title: Study on the Correlation Between MAPT Haploid H1b and the Damage of Blood-brain Barrier in Dorsal Medulla Oblongata and Autonomic Dysfunction in Parkinson's Disease
Brief Title: MAPT Haploid H1b and the Damage of BBB in Dorsal Medulla Oblongata and Autonomic Dysfunction in PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-KY-034-01
Record Dates: First submitted 2022-06-08; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; MAPT genotype; autonomic dysfunction; blood brain barrier
MeSH Terms: conditions — Parkinson Disease; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Microtubule associated protein tau (MAPT ) gene is located in 17q21.3 and contains 16 exons Due to the linkage disequilibrium inheritance of genes, MAPT mainly has two extended haplotypes (H1 and H2). This gene is responsible for encoding the neuronal microtubule associated protein tau, which is mainly distributed in the axons of neurons and plays an important role in the stability and assembly of microtubules. The gene polymorphism of MAPT is related to the clinical subtype of PD, in which MAPT H1J is related to sleep behavior disorder during rapid eye movement, while the risk of postural hypotension in H1B patients is increased by 1.72 times. The above studies suggest that the gene subtype of MAPT may be related to the occurrence and progression of early autd in PD patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD with AutD: Parkinson's disease with autonomic dysfunction
  Interventions: Other: Autonomic dysfunction
- PD without AutD: Parkinson's disease without autonomic dysfunction

INTERVENTIONS:
Other: Autonomic dysfunction — Autonomic dysfunction
  Groups: PD with AutD

SUMMARY:
This study mainly explored the relationship between the permeability of the blood-brain barrier in the dorsal medulla oblongata and autonomic dysfunction, and the relationship and mechanism of MAPT genotype on the permeability of the blood-brain barrier and the progression of autonomic dysfunction in PD patients.

DETAILED DESCRIPTION:
According to the MDS 2015 clinical diagnostic criteria for Parkinson's disease and the diagnostic criteria for autonomic dysfunction (AutD), the patients were divided into PD with AutD group and PD without AutD group. DCE results, pet-pdrp+18f-dopa data and clinical evaluation (SCOPA-AUT, HRV and sleep EEG) were analyzed; Blood samples were collected to detect MAPT gene polymorphism, oligomers and phosphorylated synuclein. To explore the relationship between the permeability of the blood-brain barrier in the dorsal medulla oblongata and autonomic dysfunction, and the relationship and mechanism of MAPT genotype on the permeability of the blood-brain barrier and the progression of autonomic dysfunction in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for idiopathic PD of MDS 2015
* Age ≥ 45 years old
* Be able to complete various clinical evaluations and scales; Willing to participate in MRI, no contrast agent allergy

Exclusion Criteria:

* Dementia was diagnosed before or 1 year after the onset of motor symptoms
* Single gene form of PD
* Coexisting neuropathological diagnosis considered to affect PD progression
* Known complications affecting BBB (severe infection, cerebral infarction, etc.
* Such as comorbidities known to affect the autonomic nervous system (e.g., diabetes gangliopathy or neuropathy)
* Disturbance of consciousness, serious cerebral hemorrhage or cerebral thrombosis, serious brain tumor or brain surgery history, serious mental illness or other serious nervous system diseases, which are enough to seriously interfere with the subjects' motor and non motor symptoms
* According to the judgment of the researcher, the researcher is unable to complete the research test according to the requirements of the research scheme.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
MAPT genotype | baseline
  MAPT mainly has two extended haplotypes (H1 and H2) .
Dynamic changes of the permeability of blood-brain barrier in dorsal medulla oblongata | baseline,the sixth month,1year
  Dynamic contrast-enhanced MRI is used to measure the permeability of blood-brain barrier in dorsal medulla oblongata.Dynamic contrast ⁃ enhanced (DCE) ⁃ MRI is a very valuable quantitative MRI technology, which plays a great role in clinical research. Quantitative analysis can calculate the contrast agent concentration in the region of interest, and then improve the comparability of different research results. The permeability of blood-brain barrier is calculated by the volume transfer constant (Ktrans) between plasma and extravascular-extracellular space.
Dynamic changes of SCOPA-AUT scale | baseline,the sixth month,1 year
  The Scales for Outcomes in Parkinson's Disease-Autonomic (SCOPA-AUT) is used to evaluate autonomic nerve dysfunction. The SCOPA-AUT consists of 25 items assessing the following regions: gastrointestinal (7), urinary (6), cardiovascular (3), thermoregulatory (4), pupillomotor (1), and sexual (2 items for men and 2 items for women) dysfunction.Higher scores mean more severe autonomic dysfunction, with a minimum score of 0 and a maximum of 69.

CONTACTS AND LOCATIONS:
Overall Officials: shuzhen zhu, doctor, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China